CLINICAL TRIAL: NCT04514250
Title: Stress Aortic Valve Index for Assessing Risk in Aortic Valve Stenosis Patients
Acronym: SAVI-AoS
Status: Active, not recruiting | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, dr Pim A.L. Tonino, dr., Catharina Ziekenhuis Eindhoven
Other Study IDs: SAVI-AoS NL74875.100.20
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Discrepancies exist among aortic stenosis severity classification, patient symptom burden, and - in some cases - even survival. The new Stress Aortic Valve Index (SAVI) metric correlates better with transvalvular flow and might be a better predictor of symptoms and prognosis.

The current study will demonstrate the value of SAVI (both non-invasive and invasive) in patients with moderate aortic stenosis.

The population will consist of subjects at least 50 years old with moderate aortic stenosis (defined as aortic valve area >1.0 cm2 plus either maximal velocity 2.5-3.9 m/s or mean gradient 15-39 mmHg). Subjects with severe concomitant valve disease or severe unrevascularized coronary artery disease will be excluded, so that the isolated prognosis of aortic stenosis can be investigated.

All subjects will undergo invasive SAVI measurements during catheterization. Furthermore patients will receive non-invasive testing with an exercise echocardiogram and computed tomography (CT) scan for non-invasive SAVI measurements.

The short-term objective will compare SAVI with standard resting indexes for symptom burden, functional capacity, and biomarkers. The long-term objective will associate SAVI and standard resting indexes with clinical outcomes related to valvular disease. The investigators hypothesize that low SAVI (more marked AS during stress) will track with more symptoms and a worse prognosis.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The patients will have several study visits. The index visit will be planned to obtain informed consent and baseline parameters. The measurement visit(s) will consist of the invasive SAVI measurement, echocardiogram, stress echo imaging, 6-minute walk test, quality of life questionnaire, and the cardiac CT. During the final visit after 12 months, subjects will undergo a CT valvular calcium scan, quality of life questionnaire, and 6-minute walk test. Every subject will have an echocardiogram yearly as suggested by guideline criteria and could possibly be contacted until five years after enrollment. Blood samples will be drawn at baseline and the 1-year follow-up. Potentially the new SAVI metric could identify patients at higher risk among those with moderate gradient AS. However, since no outcome data currently exists regarding SAVI and prognosis, no conclusions could be derived from these measurements until study completion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Moderate aortic stenosis confirmed in the past 3 months by standard echocardiographic evaluation: aortic valve area >1.0 cm2 plus either maximal velocity 2.5-3.9 m/s or mean gradient 15-39 mmHg
* Ability to undergo exercise stress testing
* Ability to understand and the willingness to provide written informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study

* Any hemodynamic criterion for severe AS: maximal velocity >= 4 m/s, mean gradient >= 40mmHg, aortic valve area =< 1 cm2
* Percutaneous coronary intervention or coronary artery bypass grafting in the past three months, or have revascularization planned in the near future
* Known, unrevascularized, and severe coronary artery disease (for example a 90% diameter stenosis or FFR<0.7 in the proximal left anterior descending artery)
* Impaired left ventricular function (ejection fraction <50%)
* Unicuspid, bicuspid, or non-calcified aortic valve observed during echocardiography (note that later cusp fusion noted during study-related cardiac imaging will not exclude a subject)
* Severe aortic regurgitation, mitral valve disease, tricuspid regurgitation, or a significant intracardiac shunt
* Co-existing hypertrophic cardiomyopathy or severe septal hypertrophy >15mm
* Persistent atrial fibrillation with uncontrolled ventricular response
* Recent (within 6 weeks) acute coronary syndrome
* Estimated glomerular filtration rate ≤30 mL/min or end-stage renal disease on replacement therapy (dialysis)
* Severe COPD GOLD stage 3 or 4, home oxygen dependence, or ≥2 pulmonary inhalers (note that well-treated and stable asthma and GOLD stage 1 or 2 COPD is permitted)
* Severe comorbid condition with life expectancy <2 years
* Prior adverse reaction to dobutamine
* Severe iodine contrast allergy
* Pregnancy
* Severe pulmonary hypertension with systolic pulmonary artery pressure greater than 50mmHg or isolated and symptomatic right ventricular failure

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of symptomatic moderate aortic stenosis patients defined as: aortic valve area >1.0 cm2 plus either maximal velocity 2.5-3.9 m/s or mean gradient 15-39 mmHg. Earlier studies show that patients with moderate AS are about 75 years old and almost half are female. Their survival at one and five years is around 90% and 75% - almost the same as patients diagnosed with severe AS.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the valve metrics vs baseline clinical parameters (KCCQ) | 1 to 5 years
  A primary endpoint is the comparison of baseline clinical parameters (quality of life survey (Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS) (score 1-100), between SAVI (dimensionless) and each of mean aortic gradient (mmHg), aortic valve area (cm2), and maximal aortic valve velocity (m/s)
Evaluation of the valve metrics vs baseline clinical parameters (6MWT) | 1 to 5 years
  A primary endpoint is the comparison of baseline clinical parameters (6 minute walking test (6MWT) (meters), between SAVI (dimensionless) and each of mean aortic gradient (mmHg), aortic valve area (cm2), and maximal aortic valve velocity (m/s)
Evaluation of the valve metrics vs baseline clinical parameters (biomarkers) | 1 to 5 years
  A primary endpoint is the comparison of baseline clinical parameters (biomarkers (NT-proBNP (pg/ml); troponin (ng/L))), between SAVI (dimensionless) and each of mean aortic gradient (mmHg), aortic valve area (cm2), and maximal aortic valve velocity (m/s)

SECONDARY OUTCOMES:
Correlation between invasive (cardiac catherization) and non-invasive (stress echocardiography; computational fluid dynamics obtained from CT scan data) SAVI measurements | 1 year
  Secondary endpoints will include correlations between invasive (with pressures (mmHg) obtained during cardiac catheterization) and noninvasive (calculated based on pressures (mmHg) achieved during echocardiographic/computional fluid dynamics) SAVI (dimensionless) measurements to explore if stress assessment of the aortic valve can be imaged non-invasively or if it requires invasive hemodynamic measurement for acceptable precision. The same will be done with the cardiac CT scans that will be analyzed to see if computational fluid dynamics can simulate invasive SAVI (dimensionless).
SAVI vs. clinical outcome (number of hospitalizations (hear failure/angina/syncope/rhythm disturbances/valvular intervention/any death/cardiac death) | 1 to 5 years
  Compare SAVI (dimensionless) against standard indexes of aortic stenosis for a composite clinical endpoint of hospital admission for heart failure, angina or syncope, arrhythmia (atrial fibrillation, ventricular tachycardia), valvular intervention (SAVR, TAVI, balloon valvuloplasty), death of any cause, and cardiac death

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - UMass Medical Memorial Center, Worcester, Massachusetts
  - UTHealth Houston, McGovern Medical School, Houston, Texas
- Aalborg University Hospital, Aalborg, Denmark
- Netherlands (2):
  - Catharina Hospital Eindhoven, Eindhoven
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided